CLINICAL TRIAL: NCT02401503
Title: A Prospective, Open-label, Multicenter Phase-II Trial to Evaluate the Efficacy and Safety of a Sequential Regimen of Bendamustine Followed by GA101 and ABT-199 Followed by ABT-199 and GA101 Maintenance in CLL Patients
Brief Title: Sequential Regimen of Bendamustine-Debulking Followed by ABT-199 and GA101-Induction and -Maintenance in CLL (CLL2-BAG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Hoffmann-La Roche (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2-BAG; 2014-000580-40 (EudraCT Number)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphocytic Leucemia
Keywords: CLL
MeSH Terms: interventions — Bendamustine Hydrochloride; obinutuzumab; venetoclax

STUDY DESIGN:
Intervention Model Description: Initial treatment: 66 patients Re-treatment: 7 patients (of the initial cohort)
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine + GA101 + ABT-199 (Experimental): Bendamustine: 70mg/m² i.v. GA101: 1000 mg i.v. ABT-199: 20 - 400 mg p.o.
  Possible Re-treatment of the included patients with GA101: 1000 mg i.v. and ABT-199: 20 - 400 mg p.o.
  Interventions: Drug: Bendamustine; Drug: GA101; Drug: ABT-199

INTERVENTIONS:
Drug: Bendamustine — Debulking: Cycles 1-2, d1 & 2: 70mg/m² i.v.
Drug: GA101 — Induction: Cycle 1: d1: 100mg, d1(or 2): 900mg, d8 & 15: 1000mg; Cycle 2-6: d1: 1000mg Maintenance: Cycles 1-8 (Duration 12 weeks): d1: 1000mg
  Other Names: Obinutuzumab
Drug: ABT-199 — Induction: Cycle 2: d1-7: 20mg, d8-14: 50mg, d15-21: 100mg, d22-28: 200mg; Cycle 3-6: d1-28: 400mg Maintenance: Cycles 1-8 (Duration 12 weeks): d1-84: 400mg
  Other Names: Venetoclax, GDC-0199

SUMMARY:
The CLL2-BAG-trial is a prospective, open-label, multicenter phase-II trial to evaluate the efficacy and safety of a sequential regimen of a debulking with Bendamustine followed by an induction with GA101 (obinutuzumab) and ABT-199 (venetoclax, GDC-0199) followed by ABT-199 and GA101-maintenance in CLL patients

DETAILED DESCRIPTION:
In the CLL2-BAG-trial, a total of 62 patients of an allcomer CLL population (irrespective of physical fitness, previous therapies and prognostic factors) with an indication for treatment will be included. Patient will receive 2 cycles of debulking treatment with Bendamustine unless contraindications (e.g. refractoriness) are present or a debulking is not indicated due to a low tumor load. Afterwards, 6 cycles of induction treatment with GA101 (obinutuzumab, 3 doses in the first cycle and monthly in cycles 2-6) and ABT-199 (venetoclax, continuously starting in cycle 2 with a low dose escalation) will be applied. The primary endpoint overall response rate will be assessed at final restaging (2 months after end of induction treatment). Patients benefitting from treatment receive further therapy with GA101 (3 monthly) and ABT-199 (continuously) in a maintenance phase for up to 24 months. Maintenance treatment will be stopped in case of achievement of a complete remission and confirmation of MRD (minimal residual disease) negativity in peripheral blood or if unacceptable toxicity or progression occurs.

Since the results of the primary endpoint analysis of the CLL2-BAG trial were very promising and this trial is one of the first studies evaluating the combination of venetoclax and obinutuzumab, it is scientifically very important to follow these first patients treated with this combination as long as possible. Therefore, with amendment 4 and 5, an extended follow-up for all patients willing to continue their study participation was implemented as well as the possibility of a re-treatment with venetoclax and obinutuzumab (but without a prior bendamustine debulking) in case of a progression.

ELIGIBILITY:
Inclusion Criteria:

* documented chronic lymphocytic leukemia (CLL) requiring treatment according to International Working Group on CLL (iwCLL) criteria
* adequate renal function: a creatinine clearance ≥30ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured with 24 hr. urine collection
* adequate hematologic function: platelets ≥ 25.000/µl, neutrophils ≥ 1.000/µl and hemoglobin ≥8.0 g/dL, unless directly attributable to the patient´s CLL (e.g. bone marrow infiltration)
* adequate liver function: total bilirubin ≤2x, aspartate aminotransferase (AST) / alanin aminotransferase (ALT) ≤2.5x the institutional upper Limit of normal (ULN) value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
* negative serological testing for hepatitis B, negative testing for hepatitis-C RNA and negative HIV test within 6 weeks prior to registration
* age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2, ECOG 3 is only permitted if related to CLL
* life expectancy ≥ 6 months
* ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* transformation of CLL (i.e. Richter's transformation, prolymphocytic leukemia)
* known central nervous system (CNS) involvement
* confirmed progressive multifocal leukoencephalopathy (PML)
* malignancies other than CLL currently requiring systemic therapies
* uncontrolled infection requiring systemic treatment
* any comorbidity or organ system impairment rated with a cumulative illness rating scale (CIRS) score of 4, excluding the eyes/ears/nose/throat/larynx organ system or any other life-threatening illness, medical condition or organ system dysfunction that - in the investigator´s opinion - could compromise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g, inability to swallow tablets or impaired resorption in the gastrointestinal tract)
* requirement of therapy with strong cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors/inducers or anticoagulant with warfarin, phenprocoumon (marcumar) or other vitamin K-antagonists
* use of investigational agents within 28 days prior to registration
* known hypersensitivity to GA101 (obinutuzumab), ABT-199 (venetoclax, GDC-0199) or any of the excipients
* pregnant women and nursing mothers
* fertile men or women of childbearing potential unless surgically sterile or ≥ 2 years after the onset of menopause, or willing to use two methods of reliable contraception including one highly effective (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after end of study treatment
* vaccination with a live vaccine ≤28 days prior to registration
* legal incapacity
* prisoners or subjects who are institutionalized by regulatory or court order
* persons who are in dependence to the sponsor or an investigator

Inclusion/Exclusion criteria for extended follow-up and re-treatment

* Patients must have participated in the CLL2-BAG trial and must have benefitted from study treatment
* Only patients with a confirmed progression of CLL who are in need of treatment according to iwCLL 2008 criteria are eligible for retreatment with venetoclax and obinutuzumab
* Patients who received any subsequent treatment for CLL outside the study are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 84 days after start of the last cycle of induction therapy
  Proportion of patients responding according to international working Group on chronic lymphocytic leukemia criteria

SECONDARY OUTCOMES:
Adverse Events (AEs) and adverse events of special interest (AESI) | up to 40 months after first dose of study drug
  Type, frequency and severity of adverse events (AEs) and adverse events of special interest (AESI) and their relationship to study treatment
Rate of minimal residual disease (MRD) | up to 40 months
  Rate of MRD responses in peripheral blood measured by immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Paula Cramer, Dr. med., Principal Investigator — German CLL Study Group
Locations (1):
- German CLL Study Group, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cramer P, Tausch E, von Tresckow J, Giza A, Robrecht S, Schneider C, Furstenau M, Langerbeins P, Al-Sawaf O, Pelzer BW, Fink AM, Fischer K, Wendtner CM, Eichhorst B, Kneba M, Stilgenbauer S, Hallek M. Durable remissions following combined targeted therapy in patients with CLL harboring TP53 deletions and/or mutations. Blood. 2021 Nov 11;138(19):1805-1816. doi: 10.1182/blood.2020010484. PMID 34086865
- [Background] Cramer P, von Tresckow J, Bahlo J, Robrecht S, Langerbeins P, Al-Sawaf O, Engelke A, Fink AM, Fischer K, Tausch E, Seiler T, Fischer von Weikersthal L, Hebart H, Kreuzer KA, Bottcher S, Ritgen M, Kneba M, Wendtner CM, Stilgenbauer S, Eichhorst B, Hallek M. Bendamustine followed by obinutuzumab and venetoclax in chronic lymphocytic leukaemia (CLL2-BAG): primary endpoint analysis of a multicentre, open-label, phase 2 trial. Lancet Oncol. 2018 Sep;19(9):1215-1228. doi: 10.1016/S1470-2045(18)30414-5. Epub 2018 Aug 13. PMID 30115596
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- See also: Click here for more information about this study: CLL2-BAG (German CLL Study Group) — https://www.dcllsg.com/cll2-bag/